CLINICAL TRIAL: NCT00285025
Title: A Phase II, Multicenter, Multinational, Randomized, Double-Blind, Placebo-Controlled, Efficacy, Safety and Tolerability Study of SR57667B in Patients With Mild-to-Moderate Alzheimer's Disease
Brief Title: Study of the Effect of SR57667B in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5286; SR57667B
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2006-02-01 (Estimated); Status verified 2006-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; nerve growth factors; Clinical Trial
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: SR57667B

SUMMARY:
The primary objective is to demonstrate that SR57667B at the dose of 4 mg/day, in comparison to placebo, decreases the decline in cognitive performance and the global clinical decline over 1 year in patients with mild to moderate AD.

Secondary objectives are to assess the effect of SR57667B on functional decline and its safety/tolerability in patients with mild to moderate AD, and to document plasma concentrations of SR57667 in patients with mild to moderate AD.

DETAILED DESCRIPTION:
Multinational, multicenter, randomized, parallel-group, double-blind, phase II study

ELIGIBILITY:
Inclusion Criteria:

* Male / female outpatients.
* Age > 50 years at screening.
* Dementia of Alzheimer's Type (DSM-IV 290.0) according to DSM-IV criteria, Probable AD according to NINCDS-ADRDA criteria, Mini-Mental State Examination score > 12 and < 26.
* Untreated or treated for a minimum of 6 months before randomization with a stable dose of the cholinesterase inhibitors
* Generally healthy and ambulatory or ambulatory-aided (i.e., walker or cane).
* Presence of a reliable caregiver.
* Patient, identified caregiver and, if applicable, patient surrogate (primary relative, legal guardian, medical proxy) have given their informed written consent and are capable of following study procedures

Exclusion Criteria:

* Any cause of dementia not due to Alzheimer's disease, Delusions, delirium, psychosis, depression, or other significant psychiatric disorder.
* Treatment with any registered or putative cognitive enhancer or disease modifier other than donepezil, rivastigmine or galantamine.
* Females who are pregnant or breast-feeding. Females of child bearing potential (premenopausal female biologically capable of becoming pregnant) must have a confirmed negative serum b-HCG pregnancy test at the screening visit, and must use an acceptable method of birth control.
* Severe or unstable cardiovascular, respiratory, renal, hematological, endocrinological, neurological or other somatic disease.
* Use of CYP3A4 strong inhibitors
* Evidence (detected by history, physical examination and / or laboratory / ECG tests) of any clinically significant or unstable medical disorder that could interfere with the subject's participation in the clinical trial; interfere with the absorption, metabolism or excretion of the study medication; or interfere with the evaluation of the study drug. Alterations of laboratory tests or ECG findings of potential clinical significance.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-03; Study Completion 2005-09

PRIMARY OUTCOMES:
ADAS-cog, CDR measured at baseline and at 2, 6, 9 and 12 months.

SECONDARY OUTCOMES:
MMSE, CGIC, ADCS-ADL, NPI measured at baseline and at 2, 6, 9 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Serge GAUTHIER, MD, Study Chair — Scientific Advisory Committee; Jean-Marc ORGOGOZO, MD, Study Chair — Scientific Advisory Committee; Philip SCHELTENS, MD, Study Chair — Scientific Advisory Committee; Bengt WINBLAD, MD, Study Chair — Scientific Advisory Committee

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com